CLINICAL TRIAL: NCT06952452
Title: Multicentre, Randomised, Double-blind, Parallel-group, Phase III Study to Evaluate the Genetic Polymorphism Influence in the Response to Ranibizumab and Bevacizumab Treatment in Patients With Age-Associated Macular Degeneration.
Brief Title: Pharmacogenomics of antiVEGF in Patients With Age-Associated Macular Degeneration (AMD)
Acronym: AMD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICI21/00025; 2019-003204-12 (EudraCT Number)
Record Dates: First submitted 2024-10-28; First posted 2025-04-30 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Wet Age-related Macular Degeneration
Keywords: wAMD; antiVEGF; BVZ; RBZ; AMD; pharmacogenomics
MeSH Terms: interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 into one of two treatment arms: ranibizumab or bevacizumab. Patients who meet elegibility criteria and decline participation due to treatment randomization, will participate in an observational follow-up.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bevacizumab, BVZ (group A) (Experimental): A cycle of 3 intravitreal injections every 4-6 weeks of BVZ
  Interventions: Drug: Bevacizumab
- Ranibizumab, RBZ (group B) (Active Comparator): A cycle of 3 intravitreal injections every 4-6 weeks of RBZ
  Interventions: Drug: Ranibizumab Ophthalmic

INTERVENTIONS:
Drug: Bevacizumab — The dosage for each intravitreal injection is 1.25mg of BVZ in 0.05ml
  Other Names: Avastin; L01XC07
  Arms: Bevacizumab, BVZ (group A)
Drug: Ranibizumab Ophthalmic — The dosage for each intravitreal injection contains 0.5mg of RBZ in 0.05ml
  Other Names: Lucentis; S01LA04
  Arms: Ranibizumab, RBZ (group B)

SUMMARY:
This is a phase III, multicenter, randomized double-blinded clinical trial with two parallel groups (ranibizumab and bevacizumab) and an observational follow-up of patients who meet elegibility criteria and decline participation due to treatment randomization. It will be performed involving 630 eyes from patients with wet age-related macular degeneration (wAMD) diagnosis without another eye disease. This clinical trial compares the treatment response for 3 years, considering genetic variants already studied between the eyes treated with one of the first options of anti-VEGF used in patients with wAMD, (ranibizumab) and the most cost-effective anti-VEGF (bevacizumab; off-label use)

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with neovascular Age-related Macular Degeneration
* Age of 50 years or older.
* That at the discretion of the ophthalmologist has an indication of receiving treatment with an anti-VEGF agent as usual in clinical practice.
* Without previous treatment in the eye under study (no previous treatment for AMD).

Exclusion Criteria:

* Participate or have participated in another clinical trial with an experimental drug in the last 6 months.
* Patients with other eye diseases, p. eg, advanced glaucoma or visually significant cataracts, which are likely to require surgery during the follow-up period in the eye under study.
* Concomitant, ocular or systemic, administration of drugs up to 3 months before the treatment with another anti-VEGF in the contralateral eye.
* High cardiovascular risk: poorly controlled arterial hypertension, history or risk of arterial thromboembolic events, history of stroke or acute myocardial infarction, anticoagulant treatment, proteinuria or major elective surgery within 3 months.
* Ophthalmological risk with the intraocular injection (all intravitreal treatments): active or suspected ocular or periocular infection, severe blepharitis, history of endophthalmitis, history of retinal detachment, myopathy, glaucoma.
* Hypersensitivity to the active substance or to the excipients.
* Diabetic retinopathy documented.
* Pregnant or nursing (lactating) women.

Patients who meet elegibility criteria and decline participation due to treatment randomization, will participate in an observational follow-up, collecting saliva for the analysis of genetic polymorphisms and clinical data related to antiVEGF received out of the clinical trial and AV, OCT results and adverse events registered in medical records at 6m, 12m, 24m, 36m.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Frequency of Genetic Polymorphism in VEGFA Associated With Anti-VEGF Treatment Response in AMD Patients | From baseline, first dose, up to 3 years
  Proportion of patients carrying the VEGFA genetic polymorphism (VEGFA, CFH, CTFG, ARMS2, HTRA1, OR52B4, LOC387715, LOC100287225, LEPR, SERPINF1), as determined by genotyping of DNA extracted from saliva samples.
  This measure will be correlated with response to anti-VEGF therapy (ranibizumab or aflibercept).
  Unit of Measure: % of participants with polymorphism. Measurement Tool: Genotyping assay on saliva-derived DNA (e.g., TaqMan PCR-based method).

SECONDARY OUTCOMES:
Change in Visual Acuity Over Time in Patients With AMD Receiving Anti-VEGF Therapy | Baseline, 6 months, 12 months, 24 months, 36 months
  Visual acuity (VA), measured in number of letters read on the ETDRS chart, at baseline and at months 6, 12, 24, and 36. The change from baseline will be analyzed to assess treatment response over time.
  Unit of Measure: Number of letters (ETDRS scale). Measurement Tool: ETDRS (Early Treatment Diabetic Retinopathy Study) visual acuity chart.
Change in Retinal Fluid and Foveal Thickness Over Time as Measured by OCT in Patients With AMD Treated With Anti-VEGF Therapy | Baseline, 6 months, 12 months, 24 months, 36 months
  Retinal anatomical changes assessed by OCT, including presence and amount of intraretinal and/or subretinal fluid, and central foveal thickness (in microns), measured at baseline and at months 6, 12, 24, and 36. Differences between treatment arms (ranibizumab vs. bevacizumab) will be evaluated over time.
  Unit of Measure: Microns for foveal thickness; qualitative presence/absence or categorical grading of retinal fluid Measurement Tool: Spectral-domain Optical Coherence Tomography (SD-OCT)
Distribution of Sex Among Patients With AMD Receiving Anti-VEGF Therapy | At baseline
  Proportion of male and female participants in the study population, analyzed in relation to treatment response to anti-VEGF drugs.
  Unit of Measure: % of participants by sex. Measurement Tool: Demographic data collected via clinical records.
Distribution of Age at Diagnosis in Patients With AMD Receiving Anti-VEGF Therapy | At baseline
  Age in years at time of AMD diagnosis for each participant. Age will be analyzed as a continuous variable in relation to treatment response.
  Unit of Measure: Years. Measurement Tool: patient-reported age or medical record.
Proportion of Smokers Among Patients With AMD Receiving Anti-VEGF Therapy | At baseline
  Proportion of participants with a history of tobacco use at baseline, categorized as current, former, or never smokers.
  Unit of Measure: % of participants by smoking status. Measurement Tool: Patient-reported history via questionnaire or clinical interview.
Weight of Patients With AMD Receiving Anti-VEGF Therapy | At baseline
  Mean weight of participants measured at baseline. Weight will be used both as a descriptive baseline characteristic and as part of the BMI calculation.
  Unit of Measure: Kilograms (kg) Measurement Tool: Calibrated digital scale
Height of Patients With AMD Receiving Anti-VEGF Therapy | At baseline
  Mean height of participants measured at baseline. Height will be used both as a descriptive baseline characteristic and as part of the BMI calculation.
  Unit of Measure: Meters (m) Measurement Tool: Stadiometer
Prevalence of Obesity in Patients With AMD Receiving Anti-VEGF Therapy | At baseline
  Proportion of participants with obesity, defined as BMI ≥ 30 kg/m² at baseline. Unit of Measure: % of participants with BMI ≥ 30 kg/m². Measurement Tool: Body Mass Index (BMI) calculated from measured height and weight.
Prevalence of Hypertension in Patients With AMD Receiving Anti-VEGF Therapy | At baseline
  Proportion of participants with a diagnosis of hypertension at baseline. Unit of Measure: % of participants with hypertension. Measurement Tool: Clinical diagnosis from patient medical records or blood pressure measurement (≥140/90 mmHg).
Number of Participants With Ocular and Systemic Adverse Events Associated With Intravitreal Anti-VEGF Therapy | From intravitreal injection, up to 3 years
  Total number of participants experiencing ocular or systemic adverse events, including cardiovascular events (e.g., myocardial infarction, stroke), following intravitreal injection of ranibizumab or bevacizumab. Events will be assessed cumulatively from the third intravitreal injection through the 3-year follow-up.
  Unit of Measure: Number of participants with at least one adverse event. Measurement Tool: Clinical assessment and adverse event reporting as per standard pharmacovigilance procedures.
Total Direct Healthcare Cost per Patient for Anti-VEGF Therapy Over One Year From the Health System Perspective | From baseline up to 1 year
  Total direct healthcare cost per patient treated with ranibizumab or bevacizumab over a 1-year period, based on a cost minimization analysis assuming similar clinical efficacy. Costs will be calculated from the perspective of the Spanish National Health System (SNS) and will include drug acquisition (considering container cost and fractionation), number of intravitreal injections, pharmacogenomic testing, and clinical monitoring. The NEI VFQ-25 composite score will be used to contextualize quality-of-life outcomes within the economic evaluation.
  Unit of Measure: Euros per patient. Measurement Tool: Cost minimization analysis based on administrative and billing records; NEI VFQ-25 (National Eye Institute Visual Function Questionnaire) for quality-of-life scoring.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital la Esperanza, Barcelona
  - Unidad Central de Investigación Clínica y Ensayos Clínicos (UCICEC La Paz), Madrid

IPD SHARING:
Plan to Share IPD: Undecided